CLINICAL TRIAL: NCT07376148
Title: Fractional CO2 Laser-assisted Delivery of Hyaluronic Acid, Ascorbic Acid and Sodium DNA For Enhancing Facial Skin Quality in Individuals Over the Age of 30
Acronym: FCLADHAAASDFSQ
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2025/05/04
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Skin Quality Improvement; Photo-aged Skin; Drug Delivery Systems
Keywords: Skin Quality; Fractional Ablative Resurfacing;; Topical Drugs
MeSH Terms: interventions — Hyaluronic Acid; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The study involves the application of ascorbic acid, hyaluronic acid, and sodium DNA in preparation for their use following the administration of a fractional CO2 laser treatment. Participants will attend a total of four sessions. During the initial session, participants will complete and sign a consent form, baseline photographs will be captured for documentation purposes, and an initial assessment will be conducted using the SASSQ. At the second session, the fractional CO2 laser will be applied, followed by the application of the topical medication to the facial area. During the third and fourth sessions, scheduled one week and four weeks post-treatment, respectively, the facial dermal effects will be objectively evaluated using the SASSQ scale, and any adverse effects will be assessed and documented through photographs. To facilitate the analysis and comparison of variables, an analysis of variance will be conducted utilizing the ANOVA test for repeated measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application of ascorbic acid, hyaluronic acid, and sodium DNA in preparation for their use following (Experimental): Participants will attend a total of four sessions. During the initial session, participants will complete and sign a consent form, baseline photographs will be captured for documentation purposes, and an initial assessment will be conducted using the SASSQ. At the second session, the fractional CO2 laser will be applied, followed by the application of the topical medication to the facial area. During the third and fourth sessions, scheduled one week and four weeks post-treatment, respectively, the facial dermal effects will be objectively evaluated using the SASSQ scale, and any adverse effects will be assessed and documented through photographs.
  Interventions: Drug: topical hyaluronic acid, ascorbic acid, and sodium DNA following ablative fractional laser treatment

INTERVENTIONS:
Drug: topical hyaluronic acid, ascorbic acid, and sodium DNA following ablative fractional laser treatment — The study involves the application of ascorbic acid, hyaluronic acid, and sodium DNA in preparation for their use following the administration of a fractional CO2 laser treatment

SUMMARY:
Evaluate the effectiveness of topical hyaluronic acid, ascorbic acid, and sodium DNA following ablative fractional laser treatment in objectively reversing facial skin alterations induced by photoaging.

DETAILED DESCRIPTION:
The study involves the application of ascorbic acid, hyaluronic acid, and sodium DNA in preparation for their use following the administration of a fractional CO2 laser treatment. Participants will attend a total of four sessions. During the initial session, participants will complete and sign a consent form, baseline photographs will be captured for documentation purposes, and an initial assessment will be conducted using the SASSQ. At the second session, the fractional CO2 laser will be applied, followed by the application of the topical medication to the facial area. During the third and fourth sessions, scheduled one week and four weeks post-treatment, respectively, the facial dermal effects will be objectively evaluated using the SASSQ scale, and any adverse effects will be assessed and documented through photographs.

To facilitate the analysis and comparison of variables, an analysis of variance will be conducted utilizing the ANOVA test for repeated measures. The IBM SPSS Statistics software, version 29.0, will be employed for this purpose. A p-value of less than 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, over 30 years of age, with moderate skin changes associated with elasticity, wrinkles, roughness, pigmentation, erythema, and pore size; with at least 12 points on the SASSQ scale. Fitzpatrick skin type I-III. Participants who agree to take part in the protocol

Exclusion Criteria:

* Fitzpatrick skin type IV-VI. Local infections or inflammatory disorders.. Neoplasms suspected of being malignant. Allergy to hyaluronic acid, ascorbic acid, and sodium DNA. Hypersensitivity to fractional CO2 laser. Pregnancy or breastfeeding. Local or systemic adverse reaction

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Skin quality | From enrollment to the end of treatment at 4 weeks
  Quantitative enhancement that can be assessed using a validated scale (SASSQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología F.A.P. Conde de Valenciana, I.A.P., Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Abril 2026 - December 2026

REFERENCES:
- [Result] Kieser M, Wassmer G. On the use of the upper confidence limit for the variance from a pilot sample for sample size determination. Biom J. 1996;38(8):941-9. doi: 10.1002/bimj.4710380806
- [Result] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Result] Eiben-Nielson C, Kerscher M. Development and validation of a global photonumeric scale for evaluating skin quality of aged female facial skin. J Cosmet Dermatol. 2021 Dec;20(12):4032-4039. doi: 10.1111/jocd.14058. Epub 2021 Mar 24. PMID 33690945
- [Result] Fitzpatrick RE. Maximizing benefits and minimizing risk with CO2 laser resurfacing. Dermatol Clin. 2002 Jan;20(1):77-86. doi: 10.1016/s0733-8635(03)00047-0. PMID 11859596
- [Result] Iaconisi GN, Lunetti P, Gallo N, Cappello AR, Fiermonte G, Dolce V, Capobianco L. Hyaluronic Acid: A Powerful Biomolecule with Wide-Ranging Applications-A Comprehensive Review. Int J Mol Sci. 2023 Jun 18;24(12):10296. doi: 10.3390/ijms241210296. PMID 37373443
- [Result] Palomar-Llatas F, Castellano-Rioja E, Arantón-Areosa L, Fornes-Pujalte B, Palomar-Albert D, Díez-Fornes P, et al. Abordaje de las lesiones cutáneas más frecuentes en el envejecimiento. Enfermería Dermatológica [Internet]. 2020;14(39). doi: 10.5281/zenodo.3779297
- [Result] Holck DE, Ng JD. Facial skin rejuvenation. Curr Opin Ophthalmol. 2003 Oct;14(5):246-52. doi: 10.1097/00055735-200310000-00004. PMID 14502051
- [Result] Cafardi JA, Elmets CA. T4 endonuclease V: review and application to dermatology. Expert Opin Biol Ther. 2008 Jun;8(6):829-38. doi: 10.1517/14712598.8.6.829. PMID 18476794
- [Result] Yarosh DB, Rosenthal A, Moy R. Six critical questions for DNA repair enzymes in skincare products: a review in dialog. Clin Cosmet Investig Dermatol. 2019 Aug 29;12:617-624. doi: 10.2147/CCID.S220741. eCollection 2019. PMID 31695467
- [Result] Ge S, Chung HJ, Weiss RA. Histologic Effects of Fractional Lasers and Energy-Based Devices on Intradermally Injected Hyaluronic Acid Filler for Improving Skin Smoothness. Lasers Surg Med. 2025 Jan;57(1):96-100. doi: 10.1002/lsm.23863. Epub 2024 Nov 29. PMID 39611591
- [Result] Zhang J, Xu F, Lin H, Ma Y, Hu Y, Meng Q, Lin P, Zhang Y. Efficacy of fractional CO2 laser therapy combined with hyaluronic acid dressing for treating facial atrophic acne scars: a systematic review and meta-analysis of randomized controlled trials. Lasers Med Sci. 2023 Sep 19;38(1):214. doi: 10.1007/s10103-023-03879-y. PMID 37723352
- [Result] Weinstein-Oppenheimer CR, Brown DI, Coloma R, Morales P, Reyna-Jeldes M, Díaz MJ, Sánchez E, Acevedo CA. Design of a hybrid biomaterial for tissue engineering: Biopolymer-scaffold integrated with an autologous hydrogel carrying mesenchymal stem-cells. Mater Sci Eng C Mater Biol Appl. 2017 Oct 1;79:821-830. doi: 10.1016/j.msec.2017.05.116
- [Result] Murphy SV, Skardal A, Song L, Sutton K, Haug R, Mack DL, Jackson J, Soker S, Atala A. Solubilized Amnion Membrane Hyaluronic Acid Hydrogel Accelerates Full-Thickness Wound Healing. Stem Cells Transl Med. 2017 Nov;6(11):2020-2032. doi: 10.1002/sctm.17-0053. Epub 2017 Sep 23. PMID 28941321
- [Result] Fanian F, Deutsch JJ, Bousquet MT, Boisnic S, Andre P, Catoni I, Beilin G, Lemmel C, Taieb M, Gomel-Toledano M, Issa H, Garcia P. A hyaluronic acid-based micro-filler improves superficial wrinkles and skin quality: a randomized prospective controlled multicenter study. J Dermatolog Treat. 2023 Dec;34(1):2216323. doi: 10.1080/09546634.2023.2216323. Epub 2023 Aug 14. PMID 37577796
- [Result] Abatangelo G, Vindigni V, Avruscio G, Pandis L, Brun P. Hyaluronic Acid: Redefining Its Role. Cells. 2020 Jul 21;9(7):1743. doi: 10.3390/cells9071743. PMID 32708202
- [Result] Boo YC. Ascorbic Acid (Vitamin C) as a Cosmeceutical to Increase Dermal Collagen for Skin Antiaging Purposes: Emerging Combination Therapies. Antioxidants (Basel). 2022 Aug 26;11(9):1663. doi: 10.3390/antiox11091663. PMID 36139737
- [Result] Bhowmick S, Rother S, Zimmermann H, Lee PS, Moeller S, Schnabelrauch M, Koul V, Jordan R, Hintze V, Scharnweber D. Biomimetic electrospun scaffolds from main extracellular matrix components for skin tissue engineering application - The role of chondroitin sulfate and sulfated hyaluronan. Mater Sci Eng C Mater Biol Appl. 2017 Oct 1;79:15-22. doi: 10.1016/j.msec.2017.05.005. Epub 2017 May 4. PMID 28629001
- [Result] Njus D, Kelley PM, Tu YJ, Schlegel HB. Ascorbic acid: The chemistry underlying its antioxidant properties. Free Radic Biol Med. 2020 Nov 1;159:37-43. doi: 10.1016/j.freeradbiomed.2020.07.013. Epub 2020 Jul 30. PMID 32738399
- [Result] Waibel JS, Mi QS, Ozog D, Qu L, Zhou L, Rudnick A, Al-Niaimi F, Woodward J, Campos V, Mordon S. Laser-assisted delivery of vitamin C, vitamin E, and ferulic acid formula serum decreases fractional laser postoperative recovery by increased beta fibroblast growth factor expression. Lasers Surg Med. 2016 Mar;48(3):238-44. doi: 10.1002/lsm.22448. Epub 2015 Nov 27. PMID 26612341
- [Result] Hsiao CY, Huang CH, Hu S, Ko YS, Sung HC, Chen CC, Huang SY. Fractional carbon dioxide laser treatment to enhance skin permeation of ascorbic acid 2-glucoside with minimal skin disruption. Dermatol Surg. 2012 Aug;38(8):1284-93. doi: 10.1111/j.1524-4725.2012.02454.x. Epub 2012 Jun 5. PMID 22672633
- [Result] Farris PK. Topical vitamin C: a useful agent for treating photoaging and other dermatologic conditions. Dermatol Surg. 2005 Jul;31(7 Pt 2):814-7; discussion 818. doi: 10.1111/j.1524-4725.2005.31725. PMID 16029672
- [Result] Ibrahim O, Wenande E, Hogan S, Arndt KA, Haedersdal M, Dover JS. Challenges to laser-assisted drug delivery: Applying theory to clinical practice. Lasers Surg Med. 2018 Jan;50(1):20-27. doi: 10.1002/lsm.22769. Epub 2017 Nov 20. PMID 29154501
- [Result] Muskat A, Kost Y, Balazic E, Cohen JL, Kobets K. Laser-Assisted Drug Delivery in the Treatment of Scars, Rhytids, and Melasma: A Comprehensive Review of the Literature. Aesthet Surg J. 2023 Feb 21;43(3):NP181-NP198. doi: 10.1093/asj/sjac286. PMID 36325715
- [Result] Waibel JS, Rudnick A. Laser-assisted delivery to treat facial scars. Facial Plast Surg Clin North Am. 2017;25(1):105-17. doi: 10.1016/j.fsc.2016.08.010
- [Result] Seo HM, Choi JY, Min J, Kim WS. Carbon dioxide laser combined with botulinum toxin A for patients with periorbital syringomas. J Cosmet Laser Ther. 2016 Jun;18(3):149-53. doi: 10.3109/14764172.2015.1052517. Epub 2016 Mar 31. PMID 26073121
- [Result] Mohamed HA, Mohammed GF, Gomaa AH, Eyada MM. Carbon dioxide laser plus topical 5-fluorouracil: a new combination therapeutic modality for acral vitiligo. J Cosmet Laser Ther. 2015;17(4):216-23. doi: 10.3109/14764172.2014.1003241. Epub 2015 Jan 30. PMID 25549816
- [Result] Franz TJ. Kinetics of cutaneous drug penetration. Int J Dermatol. 1983 Nov;22(9):499-505. doi: 10.1111/j.1365-4362.1983.tb02187.x. No abstract available. PMID 6358066
- [Result] Scott JA, Banga AK. Cosmetic devices based on active transdermal technologies. Ther Deliv. 2015;6(9):1089-99. doi: 10.4155/tde.15.64. Epub 2015 Sep 21. PMID 26389853
- [Result] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Result] Alegre-Sánchez A, Jiménez-Gómez N, Boixeda P. Vehiculización de fármacos asistida por láser. Actas Dermo-sifiliográficas. 2018;109:858-867. doi: 10.1016/j.ad.2018.07.008
- [Result] Sklar LR, Burnett CT, Waibel JS, Moy RL, Ozog DM. Laser assisted drug delivery: a review of an evolving technology. Lasers Surg Med. 2014 Apr;46(4):249-62. doi: 10.1002/lsm.22227. Epub 2014 Mar 24. PMID 24664987
- [Result] Zaleski-Larsen LA, Fabi SG. Laser-Assisted Drug Delivery. Dermatol Surg. 2016 Aug;42(8):919-31. doi: 10.1097/DSS.0000000000000556. PMID 27191783
- [Result] de Szalay S, Wertz PW. Protective Barriers Provided by the Epidermis. Int J Mol Sci. 2023 Feb 5;24(4):3145. doi: 10.3390/ijms24043145. PMID 36834554